CLINICAL TRIAL: NCT00182312
Title: Efficacy and Safety of Methylxanthines in Very Low Birthweight Infants
Brief Title: Caffeine for Apnea of Prematurity (CAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CTMG-1999-CAP; ISRCTN44364365 (Registry Identifier: Current Controlled Trials); MCT-13288 (Other Grant/Funding Number: CIHR); MOP-102601 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2016-09

CONDITIONS: Apnea of Prematurity
Keywords: preterm infants; very low birthweight; apnea of prematurity; methylxanthines; developmental disabilities
MeSH Terms: conditions — Apnea; Developmental Disabilities | interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Caffeine citrate injection — Loading dose: 20 mg/kg administered over at least 30 minutes via IV infusion or over at least 10 minutes via slow IV injection.
  Daily maintenance dose (to commence at least 24 hours after loading dose): 5 mg/kg, administered over at least 10 minutes via IV infusion, or over at least 5 minutes via slow IV injection. Maintenance dose to be adjusted for body weight every 7 days. If indicated, maintenance dose may be increased to a maximum of 10 mg/kg. May be given orally once full enteral feeds are established.
  Duration of treatment: discontinue after infant has tolerated at least 5 consecutive days without positive pressure support AND when the infant is judged by the attending clinician to be no longer a candidate for methylxanthine therapy.
  Other Names: CafCit

SUMMARY:
At least 5 of every 1000 live-born babies are very premature and weigh only 500 to 1250 grams at birth. Approximately 30-40% of these high-risk infants either die or survive with lasting disabilities. The aim of this research is to reduce this heavy burden of illness. A multi-center randomized controlled trial has been designed in which 2000 very low birth weight infants will be enrolled. Our goal is to determine whether the avoidance of methylxanthine drugs will improve survival without disability to 18 months, corrected for prematurity.

Methylxanthine drugs such as caffeine are used to prevent or treat periodic breathing and breath-holding spells in premature infants. However, there is a striking lack of evidence for the long-term efficacy and safety of this therapy. Methylxanthines block a naturally occurring substance, called adenosine, which protects the brain during episodes of oxygen deficiency. Such episodes are common in infants who are treated with methylxanthines. It is possible that methylxanthines may worsen the damage caused by lack of oxygen. Therefore, this trial will clarify whether methylxanthines cause more good than harm in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* birthweight 500 to 1250 grams
* postnatal age day 1 to day 10
* infant considered a candidate for methylxanthine therapy by clinical staff

Exclusion Criteria:

* dysmorphic features or congenital malformations that adversely affect life expectancy or neurodevelopment
* unlikely to comply with long-term follow-up
* prior treatment with a methylxanthine

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 1999-10; Primary Completion 2007-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
combined rate of mortality and neurodevelopmental disability in survivors at a corrected age of 18 months. | corrected age of 18 months

SECONDARY OUTCOMES:
bronchopulmonary dysplasia | discharge home
necrotizing enterocolitis | discharge home
brain injury: intra- and periventricular hemorrhage, periventricular leucomalacia and/or ventriculomegaly | discharge home
retinopathy of prematurity | discharge home
growth failure | corrected age of 18 months
functional status at 5 years and at 11-12 years | corrected age of 5 years and chronological age of 11-12 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Schmidt, MD, Study Chair — McMaster University; Robin S Roberts, MTech, Study Director — McMaster University; Peter Davis, MD, Study Director — Royal Women's Hospital, Melbourne, Australia; Lex Doyle, MD, Study Director — Royal Women's Hospital, Melbourne, Australia; Arne Ohlsson, MD, Study Director — Mount Sinai Hospital, Canada; Alfonso Solimano, MD, Study Director — Children & Women's Health Centre of BC, Vancouver, Canada; Win Tin, MD, Study Director — James Cook University Hospital, Middlesbrough, UK; Keith J Barrington, MD, Study Director — Royal Victoria Hospital/McGill University, Montreal, Canada; Elizabeth Asztalos, MD, Study Director — Sunnybrook Health Sciences Centre, Toronto, Canada; Deborah Dewey, MD, Study Director — University of Calgary, Alberta, Canada; Ruth Grunau, MD, Study Director — University of British Columbia, Vancouver, Canada; Diane Moddemann, MD, Study Director — University of Manitoba, Winnipeg, Canada; Peter Anderson, PhD, Study Director — University of Melbourne, Australia
Locations (34):
- Brooklyn Hospital Center, Brooklyn, New York, United States
- Australia (4):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Women's & Children's Hospital, Adelaide, South Australia
  - Mercy Hospital for Women, Melbourne, Victoria
  - Royal Women's Hospital, Melbourne, Victoria
- Canada (15):
  - Foothills Hospital, Calgary, Alberta
  - Children's & Women's Health Centre of BC, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook & Women's College Health Science Centre, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- Germany (2):
  - Ludwig Maximilian University, Munich
  - University of Tuebingen, Tübingen
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Meir General Hospital, Kfar Saba
  - Kaplan Medical Center, Rehovot
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - University Hospital Maastricht, Maastricht
- Astrid Lindgren's Children's Hospital, Stockholm, Sweden
- Switzerland (3):
  - University Children's Hospital Basel, Basel
  - University Hospitals of Geneve, Geneva
  - University of Zurich, Zurich
- United Kingdom (3):
  - Royal Maternity Hospital, Belfast, Northern Ireland
  - South Cleveland Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Result] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Result] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Result] Davis PG, Schmidt B, Roberts RS, Doyle LW, Asztalos E, Haslam R, Sinha S, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine for Apnea of Prematurity trial: benefits may vary in subgroups. J Pediatr. 2010 Mar;156(3):382-7. doi: 10.1016/j.jpeds.2009.09.069. Epub 2009 Nov 18. PMID 19926098
- [Result] Schmidt B, Anderson PJ, Doyle LW, Dewey D, Grunau RE, Asztalos EV, Davis PG, Tin W, Moddemann D, Solimano A, Ohlsson A, Barrington KJ, Roberts RS; Caffeine for Apnea of Prematurity (CAP) Trial Investigators. Survival without disability to age 5 years after neonatal caffeine therapy for apnea of prematurity. JAMA. 2012 Jan 18;307(3):275-82. doi: 10.1001/jama.2011.2024. PMID 22253394
- [Result] Dukhovny D, Lorch SA, Schmidt B, Doyle LW, Kok JH, Roberts RS, Kamholz KL, Wang N, Mao W, Zupancic JA; Caffeine for Apnea of Prematurity Trial Group. Economic evaluation of caffeine for apnea of prematurity. Pediatrics. 2011 Jan;127(1):e146-55. doi: 10.1542/peds.2010-1014. Epub 2010 Dec 20. PMID 21173002
- [Result] Schmidt B, Davis PG, Asztalos EV, Solimano A, Roberts RS. Association between severe retinopathy of prematurity and nonvisual disabilities at age 5 years. JAMA. 2014 Feb 5;311(5):523-5. doi: 10.1001/jama.2013.282153. No abstract available. PMID 24496539
- [Result] Doyle LW, Schmidt B, Anderson PJ, Davis PG, Moddemann D, Grunau RE, O'Brien K, Sankaran K, Herlenius E, Roberts R; Caffeine for Apnea of Prematurity Trial investigators. Reduction in developmental coordination disorder with neonatal caffeine therapy. J Pediatr. 2014 Aug;165(2):356-359.e2. doi: 10.1016/j.jpeds.2014.04.016. Epub 2014 May 17. PMID 24840756
- [Derived] Doyle LW, Ranganathan S, Cheong JLY. Neonatal Caffeine Treatment and Respiratory Function at 11 Years in Children under 1,251 g at Birth. Am J Respir Crit Care Med. 2017 Nov 15;196(10):1318-1324. doi: 10.1164/rccm.201704-0767OC. PMID 28707987
- [Derived] Schmidt B, Roberts RS, Anderson PJ, Asztalos EV, Costantini L, Davis PG, Dewey D, D'Ilario J, Doyle LW, Grunau RE, Moddemann D, Nelson H, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity (CAP) Trial Group. Academic Performance, Motor Function, and Behavior 11 Years After Neonatal Caffeine Citrate Therapy for Apnea of Prematurity: An 11-Year Follow-up of the CAP Randomized Clinical Trial. JAMA Pediatr. 2017 Jun 1;171(6):564-572. doi: 10.1001/jamapediatrics.2017.0238. PMID 28437520
- [Derived] Synnes A, Anderson PJ, Grunau RE, Dewey D, Moddemann D, Tin W, Davis PG, Doyle LW, Foster G, Khairy M, Nwaesei C, Schmidt B; CAP Trial Investigator group. Predicting severe motor impairment in preterm children at age 5 years. Arch Dis Child. 2015 Aug;100(8):748-53. doi: 10.1136/archdischild-2014-307695. Epub 2015 Mar 17. PMID 25784749
- [Derived] Manley BJ, Roberts RS, Doyle LW, Schmidt B, Anderson PJ, Barrington KJ, Bohm B, Golan A, van Wassenaer-Leemhuis AG, Davis PG; Caffeine for Apnea of Prematurity (CAP) Trial Investigators; Caffeine for Apnea of Prematurity CAP Trial Investigators. Social variables predict gains in cognitive scores across the preschool years in children with birth weights 500 to 1250 grams. J Pediatr. 2015 Apr;166(4):870-6.e1-2. doi: 10.1016/j.jpeds.2014.12.016. Epub 2015 Jan 29. PMID 25641237